CLINICAL TRIAL: NCT04614376
Title: A Machine Learning Approach to Alzheimer's Detection From Continuous Blood Glucose Monitoring Data
Brief Title: Alzheimer's and Blood Glucose Levels
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Bio Conscious Technologies Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: BCT_AD_001
Record Dates: First submitted 2020-10-13; First posted 2020-11-04 (Actual); Last update posted 2020-11-04 (Actual); Status verified 2020-11

CONDITIONS: Mild Cognitive Impairment; Alzheimer Disease
MeSH Terms: conditions — Cognitive Dysfunction; Alzheimer Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Control Group: The control group participants have not been diagnosed with mild cognitive impairment or Alzheimer's disease within the past 5 years. There are no interventions to this group.
- Case Group: The case group participants have been diagnosed with mild cognitive impairment or Alzheimer's disease within the past 5 years. There are no interventions to this group.

SUMMARY:
The Alzheimer's and Blood Glucose Levels Study is researching the differences in blood glucose levels between people with and without Mild Cognitive Impairment or Alzheimer's disease with the aim of early detection of Alzheimer's Disease.

DETAILED DESCRIPTION:
This study will collect continuous glucose monitor (CGM) data from participants already using CGMs to better understand the relationship between Alzheimer's Disease and blood glucose levels. This study will use the " Endobits Companion " app for data collection. The Endobits Companion app is freely available for Android and iOS mobile devices, and was designed to keep track of patients diabetes management through a journal and relay this information with their CGM readings to their caring physician.

ELIGIBILITY:
Inclusion Criteria:

* For the case group: have been diagnosed with MCI or AD within the past 5 years.
* For the control group: have not been diagnosed with MCI or AD or another major dementia disease
* Currently using a continuous glucose monitor (CGM).
* Willing and able to provide informed consent, and to have their data collected through the Endobits Companion app. If the participant themself is unable to provide informed consent, it will be sought from their primary caregiver.

Exclusion Criteria:

* Patients younger than 50 years of age.
* Patients with a BMI lower than 18 or higher than 35.
* Patients with a major psychiatric illness (e.g., major depressive disorder, schizophrenia, bipolar disorder)
* Patients diagnosed with another major dementia disease, including vascular dementia, Lewy Body disease, Huntington's disease, Creutzfeldt-Jakob disease, and Parkinson's disease.

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population is drawn from older individuals (at least 50 years of age) with or without MCI or AD.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2020-11 (Estimated); Primary Completion 2021-08 (Estimated); Study Completion 2022-03 (Estimated)

PRIMARY OUTCOMES:
Blood Glucose Levels | This will be measured throughout the study which is a period of up to 90 days.
  All participants will use continuous glucose monitors for the period of the study. The primary outcome is to determine the difference in mean values, variability, and other patterns in blood glucose levels between the case and control groups. As there is no intervention in this study, the difference between the case and control group will be measured over the entire study period.

CONTACTS AND LOCATIONS:
Locations (1):
- Bio Conscious Technologies Inc., Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2020-08-27): https://cdn.clinicaltrials.gov/large-docs/76/NCT04614376/ICF_000.pdf